CLINICAL TRIAL: NCT02560688
Title: A Phase 1, Open-label, 2-period, Fixed-sequence Study to Evaluate the Safety and Tolerability of DS-1040b IV Infusion Coadministered With Clopidogrel in Healthy Subjects
Brief Title: Phase 1 Study to Evaluate the Safety and Tolerability of DS-1040b IV Infusion With Clopidogrel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DS1040-A-E106; 2015-003018-26 (EudraCT Number)
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2016-06

CONDITIONS: Drug Interaction
Keywords: drug interaction; clopidogrel; healthy subjects
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 - DS-1040b (Experimental): Single 12-hour intravenous infusion of DS-1040b (20 mg)
  Interventions: Drug: DS-1040b
- Period 2 - Clopidogrel (Other): Clopidogrel (Plavix) administered orally over 5 days (300 mg loading dose on Day 1 followed by 75 mg daily on Days 2-5)
  Interventions: Drug: Clopidogrel
- Period 2 - DS-1040b and Clopidogrel (Experimental): Concomitant administration of DS-1040b (20 mg single 12-hour intravenous infusion) and clopidogrel (single 75 mg oral dose)
  Interventions: Drug: DS-1040b; Drug: Clopidogrel

INTERVENTIONS:
Drug: DS-1040b — 20 mg single 12-hour intravenous infusion
  Arms: Period 1 - DS-1040b; Period 2 - DS-1040b and Clopidogrel
Drug: Clopidogrel — Clopidogrel (Plavix) administered orally 300 mg loading dose on Day 1 followed by 75 mg daily on Days 2-5
  Other Names: Plavix
  Arms: Period 2 - Clopidogrel; Period 2 - DS-1040b and Clopidogrel

SUMMARY:
This study is being conducted to test the hypothesis that coadministration of clopidogrel with DS-1040b will be safe and well tolerated. Subjects entering the study will initially receive a single 12 hour infusion of DS-1040b, to generate data on the effect of DS-1040b alone. After a wash-out period (to ensure that no DS-1040b is left in the blood) subjects will receive repeated clopidogrel doses over 5 days to generate data on the effect of clopidogrel alone. On the sixth day subjects will receive both DS-1040b and clopidogrel, and the effects will be compared to when the two treatments were given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of non-childbearing potential; subjects must be aged 18 years to 60 years, inclusive.
* Subjects with a body mass index (BMI) of 18 kg/m2 to 30 kg/m2, inclusive, and weighing between 50 kg and 100 kg, inclusive. BMI is calculated as weight [kg]/(height [m])*2.
* Subjects must be in good health as determined by medical history, physical examination and Screening investigations, and taking no regular medication.
* Female subjects must be of non-childbearing potential as follows:

  * Must be postmenopausal (the last menstrual period was at least 12 months before Screening, and a follicle-stimulating hormone [FSH] test at Screening confirms postmenopausal status); or
  * Must be surgically sterile having undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy and/or bilateral tubal ligation.
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication and dietary and lifestyle restrictions.
* Possessing sufficient intelligence to understand the nature of the study and any hazards of participating in it, and the ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Has given written consent to participate after reading the informed consent form (ICF), and after having the opportunity to discuss the study with the Investigator or his/her delegate.
* Have given written consent to have his/her data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings or laboratory values that could interfere with the objectives of the study or the safety of the subject.
* Presence or history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* Presence or history of severe adverse reaction to any medicine.
* Presence or history of malignant disease.
* Surgery (eg, stomach bypass) or medical condition that might affect absorption of medicines.
* Significant illness within 4 weeks before the dose of study medication.
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Participation in another clinical study with DS-1040b.
* Day-1 bleeding time greater than 10 minutes.
* Blood pressure (BP) and heart rate (HR) in semi-supine position at the Screening examination outside the ranges 90 to 140 mmHg systolic, 40 to 90 mmHg diastolic; HR 40 to 100 beats/min. A subject with vital signs outside the reference range for the population being studied may be included at the Investigator's discretion if it is unlikely to introduce additional risk factors and will not interfere with study procedures.
* Abnormal electrocardiogram ECG waveform morphology at Screening that would preclude accurate measurement of the uncorrected QT interval (QT) duration.
* QT interval for HR corrected using Fridericia's formula (QTcF) interval duration > 430 msec for men or > 450 msec for women, obtained as an average from the measurements on triplicate Screening ECGs.
* Use of any prescription medicine, over-the-counter (OTC) medications, herbal remedies (such as St John's Wort), or food known to be strong inhibitors or strong inducers of CYP enzymes during the 30 days before the dose of study medication; use of any other prescription or OTC medicine (except as permitted, including dietary supplements or herbal remedies, during the 7 days before the first dose of study medication.
* Consumption of certain foods or beverages before the dose and throughout the study period.
* Loss of more than 400 mL blood plasma, platelets or any other blood components during the 3 months before the first dose of study medication, or unwilling to abstain from doing so during the study and for 3 months after receipt of study medication.
* Abuse of drugs or alcohol in the past, or intake of more than 21 units of alcohol weekly (for males) or 14 units of alcohol weekly (for females).
* Use of tobacco products or nicotine-containing products during the 3 months before the dose of study medication.
* Male subjects not using adequate contraceptive methods. Male subjects have to agree to use contraception (condom with spermicide) in addition to having their female partner (if of childbearing potential) use another form of contraception (eg, an intrauterine device, diaphragm with spermicide, oral contraceptive, injectables, or subdermal hormonal implant) from the first dose until 4 months following the last dose administration. Also, the male subjects must not donate sperm until at least 4 months following the last dose administration.
* Evidence of acute or chronic infectious disease at Screening, including: positive Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) antibody, or Human Immunodeficiency Virus (HIV) antibody.
* CYP2C19 poor metabolizers.
* Subjects who have used anticoagulants (ie, warfarin, low molecular weight heparin, thrombin inhibitors), antiplatelet (eg, clopidogrel), nonsteroidal anti-inflammatory drug, and/or aspirin within 30 days prior to Period 1, Day 1.
* Subjects with a history of major bleeding or major surgical procedure of any type within 6 months before Period 1, Day 1.
* Subjects with a history of peptic ulcer, gastrointestinal bleeding including haematemesis, melena, or bleeding from haemorrhoids.
* Subjects with a history of minor bleeding episodes such as epistaxis, rectal bleeding (spots of blood on toilet paper), or gingival bleeding within 3 months before Period 1, Day 1.
* Subjects who have any family history, suspected or documented, of coagulopathy or haemoglobinopathy or evidence of abnormal coagulation parameters (eg, PT, INR or aPTT) at Screening.
* Subjects with an estimated glomerular filtration rate (eGFR) at Screening using the Modification of Diet in Renal Disease (MDRD) equation < 90 mL/min.
* Likely possibility that the subject will not cooperate with the requirements of the protocol.
* Objection by General Practitioner to subjects entering the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
number of adverse events | 5 days
  Evaluation of the safety and tolerability of DS-1040 administered alone or with clopidogrel, as determined by adverse events,from the time of dosing up to 5 days postdose.
physical exam profile | 5 days
  Evaluation of the safety and tolerability of DS-1040 administered alone or with clopidogrel, as determined by physical examination findings, vital signs, 12-lead electrocardiograms (ECGs), clinical safety laboratory tests from the time of dosing up to 5 days postdose.
bleeding time measurements | 5 days
  Evaluation of the safety and tolerability of DS-1040 administered alone or with clopidogrel, as determined by bleeding time assessments from the time of dosing up to 5 days postdose.

SECONDARY OUTCOMES:
DS-1040b plasma concentration profile Time of Maximum plasma concentration(Tmax) | 5 days
  Plasma concentrations of DS-1040 and derived PK parameters up to 5 days after a single 20 mg intravenous infusion of DS-1040 (alone and with clopidogrel).
DS-1040b plasma concentration profile Area Under the plasma concentration time Curve (AUC) | 5 days
  Plasma concentrations of DS-1040 and derived PK parameters up to 5 days after a single 20 mg intravenous infusion of DS-1040 (alone and with clopidogrel).
DS-1040b plasma concentration profile Maximum plasma concentration (Cmax) | 5 days
  Plasma concentrations of DS-1040 and derived PK parameters up to 5 days after a single 20 mg intravenous infusion of DS-1040 (alone and with clopidogrel).
changes in pharmacodynamic profile single administration | 5 days
  Change in baseline of pharmacodynamic parameters (thrombin activatable fibrinolysis inhibitor activity, clot lysis, plasma D-dimer, ADP-induced platelet aggregation) up to 5 days after a single 20 mg intravenous infusion of DS-1040 (alone and with clopidogrel).
clopidogrel plasma concentration profile Tmax | 5 days
  Plasma concentrations of Clopidogrel Active Metabolite and derived PK parameters after repeated Clopidogrel administration (alone and with DS-1040)
clopidogrel plasma concentration profile AUC | 5 days
  Plasma concentrations of Clopidogrel Active Metabolite and derived PK parameters after repeated Clopidogrel administration (alone and with DS-1040)
clopidogrel plasma concentration profile Cmax | 5 days
  Plasma concentrations of Clopidogrel Active Metabolite and derived PK parameters after repeated Clopidogrel administration (alone and with DS-1040)
changes in pharmacodynamic profile repeated administration | 5 days
  Change in baseline of pharmacodynamic parameters (thrombin activatable fibrinolysis inhibitor activity, clot lysis, plasma D-dimer, ADP-induced platelet aggregation) up to 5 days after repeated Clopidogrel administration (alone or with DS-1040)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Limsakun T, Dishy V, Mendell J, Pizzagalli F, Pav J, Kochan J, Vandell AG, Rambaran C, Kobayashi F, Orihashi Y, Warren V, McPhillips P, Zhou J. Safety and Pharmacokinetics of DS-1040 Drug-Drug Interactions With Aspirin, Clopidogrel, and Enoxaparin. J Clin Pharmacol. 2020 Jun;60(6):691-701. doi: 10.1002/jcph.1568. Epub 2020 Feb 27. PMID 32106339